CLINICAL TRIAL: NCT05472207
Title: "Multifactorial Risk Stratification in Acute and Chronic Cardiovascular Disease" ("riskINN ")
Brief Title: "Multifactorial Risk Stratification in Acute and Chronic Cardiovascular Disease"
Acronym: riskINN
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Axel Bauer, Univ.-Prof. Dr., Medical University Innsbruck
Other Study IDs: 1328/2020
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases; Healthy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cardiovascular diseases: Recording clinical data - especially risk parameters - from patients suffering from cardiovascular diseases

SUMMARY:
The aim of this study is to develop risk prediction models for the early detection of high-risk patients with structural, rhythmological or inflammatory cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Decision-eligible male and female patients ≥18 years of age
* Acute or chronic condition due to structural, rhythmologic, or inflammatory cardiovascular disease
* Informed consent for participation in the clinical trial

Exclusion Criteria:

* missing infromed consent
* pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals suffering from an acute or chronic cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
combination of cardiovascular mortality, stroke, myocardial infarction and hospitalization due to decompensated heart failure | from inclusion to end of study (max. 4 years)

SECONDARY OUTCOMES:
total mortality | from inclusion to end of study (max. 4 years)
cardiovascular mortality | from inclusion to end of study (max. 4 years)
stroke | from inclusion to end of study (max. 4 years)
myocardial infarction | from inclusion to end of study (max. 4 years)
hospitalization due to decompensated heart failure | from inclusion to end of study (max. 4 years)
hospitalization due to cardiovascular condition | from inclusion to end of study (max. 4 years)
admission to intensive care unit | from inclusion to end of study (max. 4 years)
severe arrythmic events | from inclusion to end of study (max. 4 years)

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medizinische Universität Innsbruck, Universitätsklinik für Innere Medizin III, Kardiologie & Angiologie, Innsbruck, Tyrol
  - Reha Zentrum Münster, Münster, Tyrol

IPD SHARING:
Plan to Share IPD: No